CLINICAL TRIAL: NCT05667974
Title: A Phase III, Randomized, Comparator-Controlled, Double-Blind, Multicenter Study to Evaluate the Immunogenicity, Safety and Lot to Lot Consistency of Three Lots of a PIKA Rabies Vaccine（Vero Cell）for Human Use,Freeze-dried in Healthy Adults Using a Post-Exposure Prophylaxis Schedule
Brief Title: A Study to Evaluate a PIKA Rabies Vaccine（Vero Cell）for Human Use,Freeze-dried
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yisheng Biopharma (Singapore) Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YS-002
Record Dates: First submitted 2022-12-06; First posted 2022-12-29 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2023-11

CONDITIONS: Rabies; Prevention
Keywords: Rabies; vaccine; prophylactic
MeSH Terms: conditions — Rabies | interventions — Freeze Drying

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIKA Rabies (Experimental): Receive 1 of the 3 lots of PIKA rabies vaccine via IM administration that 2-2-1 schedule with a double-dose injection on Day 0 and 3 and a single-dose injection on Day 7
  Interventions: Biological: PIKA Rabies Vaccine (Vero Cell) for Human use, Freeze-dried
- Control (Active Comparator): Receive ChiroRab via IM administration that the classic Essen 5-dose regimen 1-1-1-1-1 schedule on Days 0, 3, 7, 14 and 28
  Interventions: Biological: Chirorab

INTERVENTIONS:
Biological: PIKA Rabies Vaccine (Vero Cell) for Human use, Freeze-dried — PIKA rabies vaccine
  Arms: PIKA Rabies
Biological: Chirorab — Active Comparator
  Arms: Control

SUMMARY:
This is a phase III, randomized, comparator-controlled, double-blind, multicenter study to evaluate lot-to-lot consistency of three lots of a PIKA Rabies Vaccine, immunogenicity and safety in healthy adults using a post-exposure prophylaxis schedule. It is also the aim of this study to evaluate non-inferiority and superiority of the PIKA Rabies Vaccine compared to the rabies vaccine comparator ChiroRab.

DETAILED DESCRIPTION:
This is a phase III, randomized, comparator-controlled, double-blind, multicenter study to evaluate lot-to-lot consistency of three lots of a PIKA Rabies Vaccine, immunogenicity and safety in healthy adults using a post-exposure prophylaxis schedule. It is also the aim of this study to evaluate non-inferiority and superiority of the PIKA Rabies Vaccine compared to the rabies vaccine comparator ChiroRab.

A total of 4,500 subjects will be enrolled in the study randomized into 2:1 with 3000 subjects allocated to PIKA rabies vaccine and 1,500 allocated to receive the comparator rabies vaccine ChiroRab . There will be two study Groups: Group 1 (20%) and Group 2 (80%).

Within each study group, subjects will be randomly allocated in a 2:2:2:3 ratios to receive 1 of the 3 lots of PIKA rabies vaccine or ChiroRab. The ChiroRab group will receive the classic Essen 5 dose regimen (1-1-1-1-1 schedule on Days 0, 3, 7, 14 and 28), whilst the PIKA rabies vaccine group will receive an accelerated regimen (2-2-1 schedule with a double-dose injection on Days 0 and 3 and a single-dose injection on Day 7). For blinding purposes, normal saline will be injected on Days 14 and 28 for PIKA rabies group and Days 0 and 3 for ChiroRab group.

Group 1 will enrol a total of 900 subjects, approximately 20% of the total sample population. Subjects will be randomized at 2:2:2:3 ratio (PIKA lot #1: 200 subjects, PIKA lot #2: 200 subjects, PIKA lot #3: 200 and 300 will be randomized to receive ChiroRab). Blood will be collected pre-vaccination (Day 0) and post-vaccination on Days 7, 14, 28, 90, 180 and 365 to evaluate the primary immunogenicity, safety and secondary immunogenicity endpoints. Subjects will be followed up for the whole study period through clinic visits or phone calls.

The first 50 participants randomized in each of the 3 PIKA lots and that for the ChiroRab in Goup 1 (200 in total) will form the safety subset and will have additional blood draw for safety laboratory parameters for CBC platelet, urinalysis, serum chemistry and coagulation on Day 0 (prior to vaccination), Day 7 and Day 28.

After completion of enrolment in Group 1, Group 2 will enrol the remaining 3,600 subjects at 2:2:2:3 randomization ratio (PIKA lot #1: 800 subjects, PIKA lot #2: 800 subjects, PIKA lot #3: 800 and 1,200 will be randomized to receive ChiroRab). Blood will be collected pre-vaccination on Day 0, 7 and 365 to evaluate key secondary immunogenicity endpoints of superiority, persistence and durability of immune response as well as co-primary safety objective. Subjects will be followed up for the whole study period through clinic visits or phone calls.

After each vaccination, all subjects will be observed in the clinical site for at least 30 minutes for immediate reactions and will be followed up for solicited AEs by diary cards 7 days post each vaccination and unsolicited AEs will be collected through Day 41 post first vaccination. All subjects will be monitored for SAEs, SUSARs, AESIs, and AEs leading to study withdrawal for the whole study period.

ELIGIBILITY:
Inclusion Criteria:

* Has completed the written informed consent process.
* For Singapore sites: age ≥21 and ≤ 65 years on Study Day 0; for other country sites: age ≥18 and ≤ 65 years on Screening.
* Healthy males and females.
* No history of rabies exposure, administration of rabies vaccination or rabies immunoglobulin.
* Agree to refrain from blood donation during the course of the study.
* Be able to commit to the vaccine schedule strictly.
* Has the ability and commitment to comply with requirements of the study, such as completion of diary cards, return for follow-up visits, accessible by phone and reside within the study area for the duration of study.
* For female subjects: agree to avoid pregnancy from Study Day 0 to Study Day 90 during the course of the study. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD), or the combination of a condom or diaphragm with spermicide.

Exclusion Criteria:

* Pregnant and nursing female volunteers will be excluded from the study.
* Previous exposure to a suspect rabid animal within the last 12 months.
* Any subject who needs post-exposure prophylaxis against rabies.
* History of rabies infection or treatment (immunoglobulin or vaccine).
* History of previous rabies vaccination.
* History of hypersensitivity reaction to human immunoglobulin.
* Received any vaccine in the past 30 days before randomization except for COVID 19 and flu vaccination.
* Received immunoglobulin or blood products within 90 days before randomization or plans to receive such products at any time during active period of the study (through Day 90).
* Received any investigational therapy (including vaccine) within 90 days before randomization, or planned participation in any other investigational study during the active study period (through Day 90).
* Used immunosuppressant medications in the past 180 days (defined as more than 14 continuous days before randomization or plans to receive any products during the active vaccination period (through Day 28). An immunosuppressant dose of a glucocorticoid will be defined as a systemic dose of ≥10mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted).
* At high risk for rabies infection during the trial: (such as veterinarians and their staff, animal handlers, rabies researchers, and certain laboratory workers, persons whose activities bring them into frequent contact with rabies virus or potentially rabid bats, raccoons, skunks, cats, dogs, or other species at risk for having rabies, people travelling where rabies is enzootic, previous bite by a rabid animal with no post-exposure treatment administered).
* History of HBV or HCV infection.
* History of any past, present, or future possible immunodeficiency state including but not limited to any laboratory indication of HIV-1 infection.
* History of treatment for depression or mental illness in the past 5 years; history of any attempt of suicide.
* Bleeding disorder, or receipt of anticoagulants in the past 21 days preceding inclusion, contraindicating IM vaccination based on Investigator's judgment.
* Donation of blood within the last 2 months or who have donated plasma within the last 14 days before Study Day 0.
* Clinical signs of encephalitis.
* History or evidence on physical examination of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.
* History of neurological disorder, either congenital or acquired (e.g. seizures, meningitis, encephalitis, Guillain-Barre syndrome, dementia, vasculitis, hereditary CNS disorders).
* History of cancer (malignancy) in the past 10 years (exception is non-melanomatous skin CA).
* A history of alcohol or drug addiction in the past 2 years.
* History of hypersensitivity or serious reactions (eg. anaphylaxis, urticarial, other significant reaction) to previous vaccinations.
* Plans to permanently move from the catchment area during trial conduct.
* Concerns of compliance with protocol or social condition that makes the subject a poor candidate for the trial as determined by the PI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4500 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2025-02-21 (Estimated)

PRIMARY OUTCOMES:
Primary Immunogenicity | 14 days post-vaccination
  GMTs of rabies virus neutralizing antibodies (RVNA) at Day 14 to demonstrate lot-to-lot consistency in all subjects enrolled in Group 1
Primary Immunogenicity | 14 days post-vaccination
  RVNA seroconversion rate differences at Day 14 in all subjects enrolled in Group 1.
Co-primary Safety(solicited AEs) | 7 days after each vaccination.
  Incidence of solicited local and systemic reactions on the day of each study vaccination
Co-primary Safety(unsolicited AEs) | From day of first vaccination through 14 days after the last vaccination
  Incidence of unsolicited adverse events
Co-primary Safety(SAEs) | through study completion, an average of 1 year
  Incidence of serious adverse events (SAEs), suspected unexpected serious adverse reactions (SUSARs), adverse events of special interest (AESIs) and AEs leading to withdrawal
Co-primary Safety | through study completion, an average of 1 year
  Incidence of significant changes in the clinical laboratory test results, vital signs and physical examination by study visits.

SECONDARY OUTCOMES:
Secondary Immunogenicity | Day 28 and Day 42
  RVNA seroconversion rate differences at Day 28 and Day 42 in all subjects enrolled in Group 1
Secondary Immunogenicity | Day 7
  RVNA seroconversion rate differences at Day 7 in all subjects (Group 1 and Group 2)
Secondary Immunogenicity | Day 14, 28 and 42
  GMTs of rabies virus neutralizing antibodies (RVNA) on Day 14, 28 and 42(Group 1)
Secondary Immunogenicity | Day 90 and 180 for Group 1 only and Day 365 for all subjects (Group 1 and Group 2).
  GMTs of rabies virus neutralizing antibodies (RVNA) on Day 90 and 180 for Group 1 only and Day 365 for all subjects (Group 1 and Group 2) subjects (Group 1 and Group 2).
Secondary Immunogenicity | Day 90 and 180 for Group 1 only and Day 365 for all subjects (Group 1 and Group 2)
  RVNA seroconversion rate differences on Day 90 and 180 for Group 1 only and Day 365 for all subjects (Group 1 and Group 2)

CONTACTS AND LOCATIONS:
Locations (7):
- Pakistan (3):
  - Al-Shifa Trust Eye Hospital, Islamabad
  - Ziauddin University, Karachi
  - Central Park Teaching Hospital, Lahore
- Philippines (4):
  - TDF-Lakeview，Muntinlupa, City of Muntinlupa
  - Las Pinas Doctor's Hospital, Las Piñas
  - PGH, Manila
  - TDF - San Pablo, Laguna, San Pablo